CLINICAL TRIAL: NCT01629966
Title: A Double-blind, Placebo-Controlled Fixed-Dose Study of Vilazodone in Patients With Generalized Anxiety Disorder.
Brief Title: Safety, Efficacy and Tolerability of Vilazodone in Generalized Anxiety Disorder
Acronym: VLZ-MD-05
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VLZ-MD-05
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Results first posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-11

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; GAD
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Vilazodone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Dose-matched placebo one per day, oral administration
  Interventions: Drug: Placebo
- Vilazadone 20mg (Experimental): Vilazodone 20mg once per day, oral administration.
  Interventions: Drug: Vilazodone
- Vilazodone 40mg (Experimental): Vilazodone 40mg once per day, oral administration
  Interventions: Drug: Vilazodone

INTERVENTIONS:
Drug: Placebo — Matching 10 mg and 20 mg placebo tablets, once per day, oral administration,
  Arms: Placebo
Drug: Vilazodone — Vilazodone, 20mg, oral administration once per day.
  Arms: Vilazadone 20mg
Drug: Vilazodone — Vilazodone, 40mg, oral administration once per day.
  Arms: Vilazodone 40mg

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and tolerability of vilazodone relative to placebo in the treatment of generalized anxiety disorder (GAD)

ELIGIBILITY:
Inclusion Criteria:

* Male and female, 18 - 70 years of age
* Currently meet the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for Generalized Anxiety Disorder (GAD)
* Minimum score of 20 on the Hamilton Rating Scale for Anxiety (HAM-A)

Exclusion Criteria:

* Women who are pregnant, women who will be breastfeeding during the study and women of childbearing potential who are not practicing a reliable method of birth control
* History of meeting DSM-IV-TR criteria for any of the following:

  * Any manic or hypomanic or mixed episode, including bipolar disorder and substance-induced manic, hypomanic or mixed episode
  * Any depressive episode with psychotic or catatonic features
  * Panic disorder with or without agoraphobia
  * Obsessive-compulsive disorder
  * Schizophrenia, schizoaffective, or other psychotic disorder
  * Bulimia or anorexia nervosa
  * Presence of borderline personality disorder or antisocial personality disorder
  * Mental retardation, dementia, amnesia, or other significant cognitive disorders
* Patients who are considered a suicide risk

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2012-06-30 (Actual); Primary Completion 2014-02-28 (Actual); Study Completion 2014-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Forero, MA, Study Director — Forest Laboratories
Locations (37):
- United States (37):
  - Forest Investigative Site 001, Birmingham, Alabama
  - Forest Investigative Site 021, Beverly Hills, California
  - Forest Investigative Site 023, Glendale, California
  - Forest Investigative Site 011, Paramount, California
  - Forest Investigative Site 026, Norwich, Connecticut
  - Forest Investigative Site 027, Waterbury, Connecticut
  - Forest Investigative Site 005, Delray Beach, Florida
  - Forest Investigative Site 014, Oakland Park, Florida
  - Forest Investigative Site 019, South Miami, Florida
  - Forest Investigative Site 038, Atlanta, Georgia
  - Forest Investigative Site 035, Decatur, Georgia
  - Forest Investigative Site 028, Chicago, Illinois
  - Forest Investigative Site 030, Schaumburg, Illinois
  - Forest Investigative Site 029, Topeka, Kansas
  - Forest Investigative Site 033, Wichita, Kansas
  - Forest Investigative Site 010, Lake Charles, Louisiana
  - Forest Investigative Site 031, Baltimore, Maryland
  - Forest Investigative Site 025, Boston, Massachusetts
  - Forest Investigative Site 037, St Louis, Missouri
  - Forest Investigative Site 015, Las Vegas, Nevada
  - Forest Investigative Site 016, Berlin, New Jersey
  - Forest Investigative Site 007, Brooklyn, New York
  - Forest Investigative Site 024, New York, New York
  - Forest Investigative Site 032, New York, New York
  - Forest Investigative Site 012, New York, New York
  - Forest Investigative Site 020, Bismarck, North Dakota
  - Forest Investigative Site 008, Cincinnati, Ohio
  - Forest Investigative Site 041, Dayton, Ohio
  - Forest Investigative Site 004, Oklahoma City, Oklahoma
  - Forest Investigative Site 034, Oklahoma City, Oklahoma
  - Forest Investigative Site 013, Portland, Oregon
  - Forest Investigative Site 006, Memphis, Tennessee
  - Forest Investigative Site 017, Wichita Falls, Texas
  - Forest Investigative Site 003, Salt Lake City, Utah
  - Forest Investigative Site 018, Charlottesville, Virginia
  - Forest Investigative Site 040, Bellevue, Washington
  - Forest Investigative Site 039, Seattle, Washington

REFERENCES:
- [Derived] Khan A, Durgam S, Tang X, Ruth A, Mathews M, Gommoll CP. Post Hoc Analyses of Anxiety Measures in Adult Patients With Generalized Anxiety Disorder Treated With Vilazodone. Prim Care Companion CNS Disord. 2016 Apr 28;18(2):10.4088/PCC.15m01904. doi: 10.4088/PCC.15m01904. eCollection 2016. PMID 27486544
- [Derived] Gommoll C, Durgam S, Mathews M, Forero G, Nunez R, Tang X, Thase ME. A double-blind, randomized, placebo-controlled, fixed-dose phase III study of vilazodone in patients with generalized anxiety disorder. Depress Anxiety. 2015 Jun;32(6):451-9. doi: 10.1002/da.22365. Epub 2015 Apr 17. PMID 25891440

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Vilazadone 20mg | Vilazodone 40mg
Started | 221 | 227 | 225
Completed | 180 | 175 | 159
Not Completed | 41 | 52 | 66
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Lost to Follow-up | 10 | 13 | 9
Not completed — Withdrawal by Subject | 8 | 9 | 16
Not completed — Protocol Violation | 7 | 9 | 7
Not completed — Lack of Efficacy | 5 | 2 | 4
Not completed — Adverse Event | 11 | 18 | 30

BASELINE CHARACTERISTICS:
Population: The Safety Population consisted of all patients in the Randomized Population who took at least 1 dose of double-blind investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vilazadone 20mg | Vilazodone 40mg | Total
Number analyzed (Participants) | 221 | 227 | 225 | 673
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.0 (13.7) | 40.6 (13.7) | 39.9 (13.3) | 40.2 (13.5)
Age, Customized [Number; unit: Participants]
  < 20 | 6 | 10 | 4 | 20
  20-29 | 59 | 48 | 59 | 166
  30-39 | 50 | 54 | 50 | 154
  40-49 | 43 | 47 | 50 | 140
  50-59 | 44 | 41 | 46 | 131
  ≥ 60 | 19 | 27 | 16 | 62
Sex/Gender, Customized [Number; unit: Participants]
  Male | 78 | 78 | 83 | 239
  Female | 143 | 149 | 142 | 434
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 25 | 31 | 79
  Not Hispanic or Latino | 198 | 202 | 194 | 594
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 174 | 167 | 167 | 508
  Black or African American | 35 | 50 | 46 | 131
  Asian | 4 | 3 | 5 | 12
  American Indian or Alaska Native | 2 | 1 | 1 | 4
  Other | 6 | 6 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Hamilton Rating Scale for Anxiety (HAM-A) Total Score
Description: The Hamilton Anxiety Rating Scale (HAM-A) is a clinician-administered scale which consists of 14 items, each rated on a five point scale ranging from 0 (not present) to 4 (very severe). The highest possible score is 56, which represents the most severe form of anxiety; the lowest possible score is 0, which represents an absence of anxiety.
Time Frame: Baseline to Week 8
Population: The Intent-to-Treat (ITT) Population consisted of all patients in the Safety Population who had at least 1 postbaseline assessment of HAM-A.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Placebo | Vilazadone 20mg | Vilazodone 40mg
Number analyzed (Participants) | 221 | 223 | 223
Score on scale | 13.1 (7.93) | 12.0 (7.13) | 11.2 (7.46)
Statistical Analysis 1: Comparison: Placebo vs Vilazadone 20mg; Test type: Superiority; p = 0.0830, MMRM; Least Squares Mean Difference = -1.27, 95% CI 2-sided [-2.71 to 0.17]
Statistical Analysis 2: Comparison: Placebo vs Vilazodone 40mg; Test type: Superiority; p = 0.0156, MMRM; Least Squares Mean Difference = -1.80, 95% CI 2-sided [-3.26 to -0.34]

2. Secondary Outcome: Change From Baseline in the Sheehan Disability Scale (SDS) Total Score
Description: The Sheehan Disability Scale (SDS) is a 3-item clinician-rated questionnaire used to evaluate impairments in the domains of work, social life/leisure, and family life/home responsibility. All items are rated on an 11-point continuum (0 = no impairment to 10 = most severe) with the total SDS score ranging from 0 (no impairment) to 30 (most severe).
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on Scale
Arm/Group | Placebo | Vilazadone 20mg | Vilazodone 40mg
Number analyzed (Participants) | 221 | 223 | 223
Score on Scale | 8.4 (7.53) | 7.7 (6.51) | 6.7 (6.62)
Statistical Analysis 1: Comparison: Placebo vs Vilazadone 20mg; Test type: Superiority; p = 0.0536, MMRM; Least Squares Mean Difference = -1.37, 95% CI 2-sided [-2.75 to 0.02]
Statistical Analysis 2: Comparison: Placebo vs Vilazodone 40mg; Test type: Superiority; p = 0.0349, MMRM; Least Squares Mean Difference = -1.52, 95% CI 2-sided [-2.94 to -0.11]

ADVERSE EVENTS:
Time Frame: Adverse events were collected until week 8.
Description: The Safety Population consisted of all patients in the Randomized Population who took at least 1 dose of double-blind investigational product.
Arm/Group | Placebo | Vilazadone 20mg | Vilazodone 40mg
All-Cause Mortality (participants affected / at risk) | 0/221 | 0/227 | 0/225
Serious Adverse Events (participants affected / at risk) | 1/221 | 1/227 | 0/225
Other Adverse Events (participants affected / at risk) | 85/221 | 123/227 | 121/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=221) | Vilazadone 20mg (N=227) | Vilazodone 40mg (N=225)
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
left carpal canal hematoma (Blood and lymphatic system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=221) | Vilazadone 20mg (N=227) | Vilazodone 40mg (N=225)
Nausea (Gastrointestinal disorders) | 25 | 55 | 58
Diarrhoea (Gastrointestinal disorders) | 23 | 57 | 48
Vomiting (Gastrointestinal disorders) | 5 | 13 | 17
Dry mouth (Gastrointestinal disorders) | 12 | 10 | 10
Fatigue (General disorders) | 6 | 7 | 13
Upper respiratory tract infection (Infections and infestations) | 16 | 11 | 12
Headache (Nervous system disorders) | 18 | 32 | 25
Dizziness (Nervous system disorders) | 8 | 12 | 21
Insomnia (Psychiatric disorders) | 11 | 12 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the PI will be subject to mutual agreement between the PI and Forest Research Institute, Inc.